CLINICAL TRIAL: NCT06753448
Title: Efficacy of Diosmin and Hesperidin on Early Rehabilitation After Primary Total Knee Arthroplasty
Brief Title: Efficacy of Diosmin and Hesperidin on Early Rehabilitation After Total Knee Arthroplasty
Status: Completed | Type: Observational
Sponsor: Ankara Etlik City Hospital (Other Government)
Responsible Party: Principal Investigator, Ahmet Berkay Girgin, Principal Investigator, Ankara Etlik City Hospital
Other Study IDs: 2024-1008
Record Dates: First submitted 2024-12-18; First posted 2024-12-31 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Total Knee Arthroplasty; Venous Insufficiency of Leg
Keywords: Total knee arthroplasty; lower extremity swelling; inflammation; venous insufficiency; pain management
MeSH Terms: conditions — Inflammation; Venous Insufficiency; Agnosia | interventions — Diosmin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 14 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Study group: Participants will take diosmin and hesperidin combination in addition to standard therapy for 14 days after total knee replacement surgery.
  Interventions: Drug: Diosmin and Hesperidin Combination
- Control group: Participants will only take standard therapy for 14 days after total knee replacement surgery.

INTERVENTIONS:
Drug: Diosmin and Hesperidin Combination — Participants will take diosmin and hesperidin combination for 14 days after total knee replacement surgery.
  Groups: Study group

SUMMARY:
The goal of this clinical trial is to find out the efficacy of diosmin and hesperidin on postoperative early rehabilitation after primary total knee arthroplasty. The main questions it aims to answer are:

Does diosmin and hesperidin combined drug decreases the lower extremity swelling, pain and increases the range of motion after primary total knee arthroplasty surgery compared to standard therapy group? Does diosmin and hesperidin combined drug decreases inflammation after total knee arthroplasty surgery.

Participants will take diosmin and hesperidin in addition to standard therapy for 14 days after total knee arthroplasty surgery. Lower extremity swelling, pain and range of motion of the patients will be recorded in every visit.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent unilateral primary total knee replacement surgery
* Patients who are functionally ASA 1, ASA 2 or ASA 3.

Exclusion Criteria:

* Patients >80 years or <18 years of age
* Patients with liver insufficiency
* Patients with allergy to diosmin or hesperidin
* Patients which are not capable to communicate

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study included patients who underwent unilateral total knee arthroplasty.
Sampling Method: Probability Sample
Enrollment: 190 (Actual)
Dates: Start 2024-10-08 (Actual); Primary Completion 2025-06-10 (Actual); Study Completion 2025-06-10 (Actual)

PRIMARY OUTCOMES:
Lower extremity swelling | From enrollment to the end of the treatment at 2 weeks
  Lower extremity swelling is measured by measuring extremity diameters from 3 points (below patella, patella and above patella) and noted. Then percentage of increment or decrement of diameters is measured.

SECONDARY OUTCOMES:
Pain | From enrollment to the end of the treatment at 2 weeks
  The Visual Analog Scale is used to describe patients' pain. It is a scale that describes pain by giving numbers from 0 to 10. 0 means no pain and 10 means extreme pain.
Range of motion | From enrollment to the end of the treatment at 2 weeks
  Knee range of motion is measured with goniometer.
Blood C-reactive protein value as an inflammotory marker | From enrollment to the end of the treatment at 2 weeks
Blood erythrocyte sedimentation rate as an inflammotory marker | From enrollment to the end of the treatment at 2 weeks
Blood neutrophil/lymphocyte rate as an inflammatory marker | From enrollment to the end of the treatment at 2 weeks
Panimmune value (neutrophil x platelet x monocyte / lymphocyte) as an inflammatory marker | From enrollment to the end of the treatment at 2 weeks
The systemic immune-inflammation index (neutrophils × platelets/lymphocytes) as an inflammatory marker | From enrollment to the end of the treatment at 2 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Etlik City Hospital, Ankara, Yenimahalle, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wang Q, Jin Q, Cai L, Zhao C, Feng P, Jia J, Xu W, Qian Q, Ding Z, Xu J, Gu C, Zhang S, Shi H, Ma H, Deng Y, Zhang T, Song Y, Wang Q, Zhang Y, Zhou X, Pei L, Yang Y, Liang J, Jiang T, Li H, Liu H, Wu L, Kang P. Efficacy of Diosmin in Reducing Lower-Extremity Swelling and Pain After Total Knee Arthroplasty: A Randomized, Controlled Multicenter Trial. J Bone Joint Surg Am. 2024 Mar 20;106(6):492-500. doi: 10.2106/JBJS.23.00854. Epub 2023 Dec 18. PMID 38109425
- [Background] Fotiadis E, Kenanidis E, Samoladas E, Chytas A, Lyrtzis C, Koimtzis M, Chalidis B. Are venotonic drugs effective for decreasing acute posttraumatic oedema following ankle sprain? A prospective randomized clinical trial. Arch Orthop Trauma Surg. 2011 Mar;131(3):389-92. doi: 10.1007/s00402-011-1266-9. Epub 2011 Jan 28. PMID 21274547
- [Background] Nicolaides AN. The Benefits of Micronized Purified Flavonoid Fraction (MPFF) Throughout the Progression of Chronic Venous Disease. Adv Ther. 2020 Feb;37(Suppl 1):1-5. doi: 10.1007/s12325-019-01218-8. Epub 2020 Jan 22. PMID 31970659